CLINICAL TRIAL: NCT05888857
Title: A Multicentric Phase II Trial Evaluating MEDI5752 in Patients With Mature Tertiary Lymphoid Structures Solid Tumors.
Brief Title: MEDI5752 in Patients With Mature Tertiary Lymphoid Structures Solid Tumors.
Acronym: TAYLOR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB2023-01; 2023-503451-94 (Other: EU-CTR)
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
Keywords: tertiary lymphoid structure; solid tumor; immunotherapy
MeSH Terms: conditions — Tertiary Lymphoid Structures

STUDY DESIGN:
Intervention Model Description: 2 independent single-arm, multicenter, phase II trials, based on a two-stage three-outcome design as described in Sargent et al.
  Cohort A : patients with TLS+ IO-naïve solid tumor (miscellaneous) Cohort B: patients with TLS+ PD1/PDL1-experienced solid tumor (miscellaneous)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: patients with TLS+ IO-naïve solid tumors (Experimental): Participants with TLS+ IO-naïve solid tumors will be treated by MEDI5752
  Interventions: Drug: MEDI5752
- Cohort B: patients with TLS+ PD1/PDL1-experienced solid tumors (Experimental): Participants with TLS+ PD1/PDL1-experienced solid tumors will be treated by MEDI5752
  Interventions: Drug: MEDI5752

INTERVENTIONS:
Drug: MEDI5752 — A treatment cycle consists of 3 weeks. MEDI5752 will be administered by intravenous infusion at a fixed dose on Day 1 of each cycle

SUMMARY:
Multicentric, prospective, multi-indication, single-treatment arm, open-label phase II trial assessing the efficacy of MEDI5752

DETAILED DESCRIPTION:
Multicentric, prospective, multi-indication, single-treatment arm, open-label phase II trial assessing the efficacy of MEDI5752.

Patients with mature tertiary lymphoid structures advanced solid tumors will be included in two independent cohorts:

* Cohort A: patients with TLS+ IO-naïve solid tumor (miscellaneous)
* Cohort B: patients with TLS+ PD1/PDL1-experienced solid tumor (miscellaneous) Each cohort will rely on a two-stage three-outcome design as described in Sargent et al.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed solid tumor
2. IO-naïve patients (cohort A) OR patients with secondary resistance to PD1/PDL1 inhibitors (cohort B),
3. Patients in cohort B:

   1. have to be diagnosed previously treated with PD-L1/PD-1 inhibitors (investigational or approved),
   2. must have experienced initial clinical benefit (stable disease or better) from checkpoint inhibitor therapy for at least 4 months in which there was at least one interval scan prior to 4 months demonstrating no progression of disease.
4. Presence of mature tertiary lymphoid structures (TLS) by IHC as described in protocol section 3.2.4. Except if presence of TLS has been already confirmed by Biopathological platform at Bergonié Institute, presence of TLS should be confirmed by central review based on FFPE tumor tissue sample,
5. Advanced unresectable or metastatic solid disease,
6. Measurable disease according to RECIST v1.1
7. At least one tumor site that can be biopsied for research purpose,
8. Age ≥ 18 years,
9. Body weight > 35 kg,
10. ECOG ≤ 1,
11. Life expectancy > 3 months,
12. Adequate hematological, renal, metabolic, hepatic and cardiac functions:
13. Disease progression on prior treatment, or previously untreated disease with no available acceptable treatment. Note that no more than three lines of systemic treatment for metastatic disease are allowed and that patients with oncogenic addiction must have progressed on prior approved regimens),
14. Recovery to grade ≤ 1 from any adverse event derived from previous treatment (excluding alopecia of any grade (according to the NCI-CTCAE, version 5.0),
15. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to study entry.
16. Women and men must agree to use at least one medically highly effective method of contraception from screening, throughout the treatment period
17. Voluntary signed and dated written informed consents prior to any specific study procedure,
18. Patients with a social security in compliance with the French law.

Exclusion Criteria:

1. Any anticancer treatment within 21 days or 5 half-lives (whichever is shorter) prior to start of study treatment,
2. Whole brain radiotherapy within 14 days prior to start of study treatment,
3. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
4. Stereotactic radiosurgery within 7 days prior to start of study treatment,
5. Major surgery within 4 weeks prior to start of study treatment or still recovering from prior surgery
6. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding,
7. History of or concurrent serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study or confounds the ability to interpret data from the study
8. Prior or concurrent malignant disease
9. Any prior Grade ≥ 3 imAE while receiving immunotherapy or any unresolved imAE > Grade 1
10. For subjects who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4 : Subject must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy, must not have experienced a ≥ grade 3 imAE or an immune-related neurologic or ocular AE of any grade while receiving prior immunotherapy, must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, must not have experienced recurrence of an AE if rechallenged, and must not currently require maintenance doses of > 10 mg prednisone or equivalent per day
11. Symptomatic or actively progressing central nervous system metastases.
12. History of leptomeningeal disease or cord compression
13. Uncontrolled or symptomatic hypercalcemia
14. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiomyopathy of any etiology, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, history of myocardial infarction within the past 12 months, cardiac arrhythmia, ILD, serious chronic gastrointestinal conditions associated with diarrhea,
16. Cerebrovascular accident within 6 months prior to enrolment,
17. Any concurrent chemotherapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment.
18. Active or history of autoimmune disease immune deficiency or inflammatory disorders, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, sarcoidosis syndrome, rheumatoid arthritis, hypophysitis, uveitis, inflammatory bowel disease, diverticulitis antiphospholipid antibody syndrome, Wegener granulomatosis, Graves'disease, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis,
19. History of idiopathic pulmonary fibrosis, organizing pneumonia drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening CT scan.
20. Evidence of the following infections: active infection including tuberculosis, HIV, active hepatitis B or C or A
21. Any contraindication to biopsy for the research,
22. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
23. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons,
24. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia,
25. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment.
26. Prior allogeneic stem cell or solid organ transplantation,
27. Treatment with a live, attenuated vaccine within 30 days prior to initiation of study treatment
28. Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic Immunosuppressive medication during study treatment,
29. History of severe allergic anaphylactic reaction to chimeric or humanized antibodies or fusion proteins,
30. Known hypersensitivity to Chinese hamster ovary cell products, to any component of the MEDI5752 formulation or to any human globulin therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of the antitumor activity of MEDI5752 (independently for eah cohort) | an expected average of 6 months
  Antitumor activity will be assessed in terms of objective response rate within 24 weeks based on RECIST v1.1, independently for each cohort, and based on centralized radiological review.
  Objective response under treatment is defined as patients with confirmed complete response or confirmed partial response, as per RECIST v1.1, observed during treatment with the investigational product.
  Objective response rate is defined as the proportion of patients alive with objective response based on RECIST v1.1.
  Objective response is recorded from study treatment initiation until the end of treatment.

SECONDARY OUTCOMES:
24-weeks clinical benefit rate (CBR) independently for each cohort | 24 weeks
  CBR is defined as the proportion of patients with clinical benefit at 6 months. Clinical benefit is defined as confirmed complete response, confirmed partial response or stable disease more than 24 weeks, defined as per RECIST v1.1.
Best overall response (BoR) independently for each cohort | Throughout the treatment period, an expected average of 6 months
  BoR is defined as the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation. The best overall response is determined once all the data for the participant is known (RECIST v1.1).
Duration of response (DoR) independently for each cohort | Throughout the treatment period, an expected average of 6 months
  DoR is defined as the time from documentation of tumor response (complete response/partial response whichever is first recorded) to disease progression, according to RECIST v1.1. DoR will be assessed in responder (confirmed CR / PR) patients only.
1-year progression-free survival (PFS), independently for each cohort | 1 year
  PFS is defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause), whichever occurs first
2-year progression-free survival (PFS), independently for each cohort | 2 year
  PFS is defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause), whichever occurs first
1-year overall survival (OS), independently for each cohort | 1 year
  OS is defined as the time from study treatment initiation to death (of any cause)
2-year overall survival (OS), independently for each cohort | 2 year
  OS is defined as the time from study treatment initiation to death (of any cause)
Safety profile, independently for each cohort: Common Terminology Criteria for Adverse Events version 5 | Throughout the treatment period, an expected average of 6 months
  Number of participants with toxicity graded using the Common Terminology Criteria for Adverse Events version 5
24-weeks clinical benefit rate (iCBR) independently for each cohort as per iRECIST | 24 weeks
  iCBR is defined as the rate of patients with iCR, iPR or immune stable disease (iSD)
Duration of response (iDoR) independently for each cohort as per iRECIST | Throughout the treatment period, an expected average of 6 months
  iDoR is defined as the time from the date of the first response iCR/iPR (whichever is first recorded) to the date of PD (iUPD confirmed as iCPD) as per iRECIST. iDOR is defined for subjects with iCR or iPR. If a patient has iPR (#1) followed by a iUPD (#1) which is not confirmed, then a iPR (#2) followed by a iUPD (#2) which is confirmed at the next assessment, then the iDOR is calculated from iPR1 until iUPD2
1-year progression-free survival (iPFS), independently for each cohort as per iRECIST | 1 year
  o iPFS is defined as the time from study treatment initiation to the first occurrence of disease progression as per iRECIST or death (of any cause), whichever occurs first. The event date to be used for calculation of progression-free survival (iPFS) should be the first date at which progression criteria are met (ie, the date of iUPD) provided that iCPD is confirmed at the next assessment. If iUPD occurs, but is disregarded because of later iSD, iPR, or iCR, that iUPD date should not be used as the progression event date. If progression is not confirmed and there is no subsequent iSD, iPR, or iCR, then the iUPD date should still be used in the following scenarios: if the patient stops protocol treatment because they were not judged to be clinically stable, or no further response assessments are done (because of patient refusal, protocol noncompliance, or patient death); the next timepoint responses are all iUPD, and iCPD never occurs
2-year progression-free survival (iPFS), independently for each cohort as per iRECIST | 2 year
  o iPFS is defined as the time from study treatment initiation to the first occurrence of disease progression as per iRECIST or death (of any cause), whichever occurs first. The event date to be used for calculation of progression-free survival (iPFS) should be the first date at which progression criteria are met (ie, the date of iUPD) provided that iCPD is confirmed at the next assessment. If iUPD occurs, but is disregarded because of later iSD, iPR, or iCR, that iUPD date should not be used as the progression event date. If progression is not confirmed and there is no subsequent iSD, iPR, or iCR, then the iUPD date should still be used in the following scenarios: if the patient stops protocol treatment because they were not judged to be clinically stable, or no further response assessments are done (because of patient refusal, protocol noncompliance, or patient death); the next timepoint responses are all iUPD, and iCPD never occurs
iORR independently for each cohort | Throughout the treatment period, an expected average of 6 months
  iORR is defined as the rate of patients with immune complete or partial responses (iCR, iPR) as per iRECIST. iCR and iPR can be assigned after iUPD (immune unconfirmed progressive disease) has been documented as per iRECIST (Seymour et al)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Bergonie, Bordeaux, France